CLINICAL TRIAL: NCT07347951
Title: A Single-Center, Prospective, Phase II Clinical Study to Evaluate the Preliminary Efficacy and Safety of Short-Course Radiotherapy Followed by CAPOX Chemotherapy Combined With Serplulimab and Bevacizumab as Total Neoadjuvant Therapy for MSS-Type, Mid-Low Locally Advanced Rectal Cancer
Brief Title: A Single-center, Phase II Study on Efficacy & Safety of SCRT+CAPOX+Serplulimab+Bevacizumab for MSS Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Pan Yifei, Chief Physician, First Affiliated Hospital of Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-443
Record Dates: First submitted 2025-12-26; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: Rectal cancer; MSS; neoadjuvant immunotherapy; neoadjuvant chemoradiotherapy; Target therapy; locally advanced
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemoradiotherapy combined with ICIs and targeted therapy for MSS-type LARC (Experimental)
  Interventions: Radiation: Short-course radiotherapy; Drug: CAPOX chemotherapy; Drug: Targeted therapy with bevacizumab; Drug: Serplulimab immunotherapy

INTERVENTIONS:
Radiation: Short-course radiotherapy — Radiotherapy adopts a short-course regimen, with a dose of 5*5 Gy, administered once daily at 5 Gy per session for a total of 5 consecutive days of irradiation. It is recommended to use three-dimensional 3D-CRT or IMRT techniques. The irradiation fields include: (1) high-risk recurrence areas of the primary tumor, such as the tumor/tumor bed, mesorectal region, and presacral region. For middle and low rectal cancers, the target area should also encompass the ischioanal fossa; (2) regional lymphatic drainage areas, including the lymphatic drainage area along the common iliac vessels within the true pelvis, mesorectal region, lymphatic drainage area along the internal iliac vessels, and obturator lymph node region.
Drug: CAPOX chemotherapy — Chemotherapy with the CAPOX regimen: Capecitabine tablets are available in strengths of 0.5 g/tablet and 0.15 g/tablet; Oxaliplatin for injection is available in a strength of 0.1 g. The chemotherapy protocol is as follows: After a 7-day rest following radiotherapy, on Day 1 (D1), oxaliplatin is administered intravenously at a dose of 130 mg/m² over 2 hours; from Day 1 to Day 14 of each 3-week cycle, capecitabine is taken orally at a dose of 1000 mg/m² twice daily, with each cycle lasting 3 weeks.
Drug: Targeted therapy with bevacizumab — Targeted therapy: On Day 1 (D1) of chemotherapy initiation, bevacizumab will be administered via infusion at a dose of 7.5 mg/kg, with each treatment course lasting 3 weeks, for a total of 6 courses.
Drug: Serplulimab immunotherapy — Immunotherapy: On Day 1 (D1) of chemotherapy initiation, administer 300 mg of serplulimab, with each treatment cycle lasting 3 weeks, for a total of 6 cycles.

SUMMARY:
In a single-center, prospective, phase II study (ClinicalTrials registration number: [to be filled in]) initiated by our center to evaluate the safety and preliminary efficacy of short-course radiotherapy followed by sequential CAPOX chemotherapy combined with serplulimab and bevacizumab as total neoadjuvant therapy for MSS-type mid-low locally advanced rectal cancer, patients with mid-low MSS-type locally advanced rectal adenocarcinoma were enrolled. They received short-course radiotherapy combined with CAPEOX, serplulimab, and bevacizumab as preoperative total neoadjuvant therapy. It is anticipated that 30 subjects with locally advanced rectal cancer will be enrolled between September 2025 and September 2027.

This phase II exploratory study targets patients with locally advanced mid-low MSS/pMMR rectal cancer. It employs short-course radiotherapy combined with CAPEOX, serplulimab, and bevacizumab as preoperative total neoadjuvant therapy, aiming to clarify the efficacy and safety of this new combined radiotherapy, chemotherapy, targeted therapy, and immunotherapy approach, while also assessing the rectal/anal preservation rate and quality of life of patients. After neoadjuvant therapy, patients will undergo imaging and endoscopic evaluations to determine subsequent treatment strategies. Radical surgical resection will be performed on patients after neoadjuvant immunotherapy, followed by further analysis of the pathological complete response (pCR) rate. The primary study endpoint is the pCR rate, and secondary study endpoints include the objective response rate, organ preservation rate, 3-year disease-free survival (DFS), 3-year overall survival (OS), incidence of adverse events, and quality of life scores (EORTC QLQ-C30, EORTC QLQ-CR29, Wexner).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a desire to preserve the anus and are willing to receive the entire course of neoadjuvant therapy.

  * Aged between 18 and 75 years, with no gender restrictions.

    * Diagnosed via pelvic MRI and rectoscopy with a tumor located ≤10 cm from the anal verge, with a clinical stage of cT3-4N0/+M0, and lymph nodes confined within the mesorectum.

      * Histologically diagnosed with rectal adenocarcinoma; genetic testing indicates MSS or MSI-L, or immunohistochemistry of tumor biopsy indicates pMMR (positive for MSH1, MSH2, MSH6, and PMS2 proteins).

        * ECOG performance status score of 0-1.

          ⑥ No prior antitumor therapy, immunotherapy, anti-angiogenic therapy, or pelvic radiotherapy before inclusion.

          ⑦ Laboratory tests must meet the following criteria: i. White blood cell count ≥3.5×10⁹/L, absolute neutrophil count ≥1.8×10⁹/L, platelet count ≥100×10⁹/L, and hemoglobin ≥100 g/L; ii. INR ≤1.5, and APTT ≤1.5 times the upper limit of normal, or partial thromboplastin time (PTT) ≤1.5 times the upper limit of normal; iii. Total bilirubin ≤1.25 times the upper limit of normal; ALT and AST ≤3 times the upper limit of normal; serum albumin ≥28 g/L; iv. 24-hour creatinine clearance rate ≥50 mL/min or serum creatinine ≤1.5 times the upper limit of normal.

          ⑧ Willing to participate in this study voluntarily, sign the informed consent form, and comply with the scheduled outpatient visits and related procedural requirements to complete follow-up.

Exclusion Criteria:

* In addition to a confirmed diagnosis of rectal cancer, there is a current or past history of active malignant tumors.

  * Patients with metastases to other sites indicated by preoperative staging.

    * Patients with suspicious positive lymph nodes in non-draining areas of the rectum, such as the internal and external iliac lymph nodes, as assessed by preoperative MRI or CT.

      * Patients requiring emergency surgery due to complications such as intestinal obstruction, intestinal perforation, or intestinal hemorrhage.

        * Patients with severe comorbid conditions and an estimated life expectancy of ≤5 years.

          * Patients with known allergies to any components in the study.

            ⑦ Patients who have received immunosuppressive or systemic corticosteroid therapy for immunosuppressive purposes within 30 days prior to the initiation of study treatment.

            ⑧ Patients who have received any other investigational drug treatment (including immunotherapy) or participated in another interventional clinical trial within 30 days prior to screening.

            ⑨ Patients with other factors that may affect the study results or lead to premature termination of the study, such as alcoholism, drug abuse, other severe diseases requiring combined treatment (including psychiatric disorders), and severe laboratory abnormalities.

            ⑩ Patients with congenital or acquired immunodeficiency (such as HIV infection).

            ⑪ Vulnerable populations, including individuals with psychiatric disorders, cognitive impairments, critically ill patients, minors, pregnant women, illiterate individuals, etc.

            ⑫ Other circumstances where, in the investigator's judgment, the patient is deemed unsuitable to participate in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | After the completion of these cycles, surgical treatment will be scheduled as appropriate (within 1-2 weeks) based on the assessment results. Pathological evaluation of the postoperative specimens will be conducted according to the tumor TRG criteria.
  In tumor specimens obtained from modified neoadjuvant chemoradiotherapy combined with immunotherapy followed by TME surgical resection, no cancer cells or local lymph node metastasis of cancer cells (ypT0N0M0) are observed under a microscope.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No